CLINICAL TRIAL: NCT06276439
Title: Intraoperative Imaging of Indocyanine Green for Sentinel Lymph Node Mapping
Brief Title: Intraoperative Imaging of Lymph Nodes
Status: Recruiting | Type: Observational
Sponsor: University of Illinois at Urbana-Champaign (Other)
Collaborators: U.S. National Science Foundation (U.S. Federal Agency); Ss. Cyril and Methodius University of Skopje, Macedonia (Unknown)
Responsible Party: Sponsor
Other Study IDs: IRB23-0314
Record Dates: First submitted 2024-02-15; First posted 2024-02-26 (Actual); Last update posted 2024-02-26 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; autofluorescence; near infrared fluorescence; Indocyanine Green; ICG
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Positive lymph node detection with bioinspired sensor: We will assess the effectiveness of our bioinspired sensor in identifying affected lymph nodes in ex vivo samples. This innovative sensor integrates spectral filters and vertically aligned photodiodes, mirroring the visual capabilities of the mantis shrimp, to simultaneously capture intrinsic UV fluorescence and externally introduced NIR fluorescence from ICG.
  To minimize the potential harm from UV radiation, we employ a phased imaging approach. Initially, ICG is injected near the tumor area in the patient, utilizing its NIR fluorescence to accurately locate the lymph node and facilitate the removal of nearby fatty tissue as necessary. Following this, UV light is momentarily used to detect autofluorescence from amino acids frequently found in tumors, providing insights into the lymph node's condition. All resected samples will be analyzed by pathologist and provide ground truth.
  Interventions: Procedure: Surgical removal of breast cancer and lymph nodes
- Positive lymph node detection with highly sensitive imaging sensor: We will evaluate the performance of our sensor, characterized by low noise and high quantum efficiency, in detecting compromised lymph nodes in ex vivo samples. This advanced sensor combine spectral filters and low noise photodiodes, enabling the simultaneous detection of natural UV fluorescence and induced NIR fluorescence from ICG.
  To minimize the potential harm from UV radiation, we employ a phased imaging approach. Initially, ICG is injected near the tumor area in the patient, utilizing its NIR fluorescence to accurately locate the lymph node and facilitate the removal of nearby fatty tissue as necessary. Following this, UV light is momentarily used to detect autofluorescence from amino acids frequently found in tumors, providing insights into the lymph node's condition. All resected samples will be analyzed by pathologist and provide ground truth.
  Interventions: Procedure: Surgical removal of breast cancer and lymph nodes

INTERVENTIONS:
Procedure: Surgical removal of breast cancer and lymph nodes — The patients will undergo a surgical procedure to remove tumor tissue in the breast and its associated lymph nodes. No clinical decision is based on the imaging device tested.

SUMMARY:
One-third of the global population battles cancer, with surgery being the primary treatment for localized forms. Successful treatment often hinges on the thorough removal of primary tumors and pinpointing cancerous sentinel lymph nodes (SLN). Although modern surgical imaging and fluorescent probes enhance the detection of sentinel lymph nodes using near-infrared (NIR) fluorescence, their inability to precisely determine the nodes' status can result in additional surgeries, lymphedema, and a reduced quality of life for patients. Our research direction aims to harness the potential of bioinspired imaging technologies with the goal of precisely identifying SLN status and ensuring only the cancerous lymph nodes are excised during the initial procedure. To realize this objective, we're drawing inspiration from the mantis shrimp's visual system to create a single-chip multispectral camera that spans the deep ultraviolet to the near-infrared spectrum. Our pioneering sensor seamlessly combines perovskite nanocrystals, optical filters, and vertically-aligned photodetectors on a single chip, enabling concurrent imaging of external NIR fluorophores and internal UV fluorescence from tumor-specific markers.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the sensitivity of our two new imaging technologies (bioinspired imaging sensor and low noise imaging sensor) to detect positive sentinel lymph nodes in patients with breast cancer. We will achieve this by recording fluorescence emitted by an FDA-approved fluorescent probe known as Indocyanine Green (ICG) in ex vivo resected samples. ICG is routinely used during cancer surgeries around the world because it passively accumulates in sentinel lymph nodes. Due to the bright green coloration of ICG, surgeons can visually identify the location of the sentinel lymph node, resect them and stage the patient's cancer based on pathology results. Since ICG is also fluorescent in the near infrared spectrum, our imaging sensor can locate the sentinel lymph node quicker and more accurately than when using unaided visual inspection. Once the lymph node is located using near-infrared (NIR) imaging with indocyanine green (ICG), the extracted samples will be placed on a separate table. These samples will be subjected to ultraviolet (UV) light to check for any natural autofluorescence. A strong autofluorescence indicates the sample is likely positive or metastatic, suggesting the presence of cancer cells. Subsequent histopathological analysis will further examine these samples. The findings will be used to construct a receiver operating curve, which will help in determining the accuracy of detecting cancer-positive lymph nodes using both exogenous (ICG-induced) and endogenous (natural) fluorescence with the two imaging systems.

ELIGIBILITY:
Inclusion Criteria:

* early or progressive stage of breast cancer who needs to be treated with breast surgery

Exclusion Criteria:

* pregnant women
* previous breast cancer surgery
* history of allergic reactions to iodide or seafood allergy.
* man

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population we are studying has been diagnosed with early or progressive stage of breast cancer who need to be treated with breast surgery. The participants will undergo breast tumor removal per standard practices.
Sampling Method: Non-Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2024-02-19 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2026-02-19 (Estimated)

PRIMARY OUTCOMES:
Positive lymph node detection with custom sensors | The sample removed from the patient will be promptly imaged using our sensor, with the imaging process expected to last between 3 to 5 minutes for each sample.
  This study aims to determine the accuracy and reliability of our novel imaging technologies in identifying cancer-affected sentinel lymph nodes in breast cancer patients. Initially, we will utilize the NIR fluorescence from ICG to identify the location of lymph nodes in resected ex vivo samples. Following this, the identified lymph nodes will be exposed to UV light to detect any inherent autofluorescence. Once the imaging study is completed, a pathologist will examine all the surgically removed samples to determine whether there is metastasis in the lymph nodes, thereby establishing the definitive diagnosis.

CONTACTS AND LOCATIONS:
Overall Officials: Viktor Gruev, PhD, Principal Investigator — University of Illinois Urbana Champaign
Locations (1):
- University Clinic Hospital, Skopje, North Macedonia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Blair S, Garcia M, Davis T, Zhu Z, Liang Z, Konopka C, Kauffman K, Colanceski R, Ferati I, Kondov B, Stojanoski S, Todorovska MB, Dimitrovska NT, Jakupi N, Miladinova D, Petrusevska G, Kondov G, Dobrucki WL, Nie S, Gruev V. Hexachromatic bioinspired camera for image-guided cancer surgery. Sci Transl Med. 2021 May 5;13(592):eaaw7067. doi: 10.1126/scitranslmed.aaw7067. PMID 33952675
- [Background] Chen C, Wang Z, Wu J, Deng Z, Zhang T, Zhu Z, Jin Y, Lew B, Srivastava I, Liang Z, Nie S, Gruev V. Bioinspired, vertically stacked, and perovskite nanocrystal-enhanced CMOS imaging sensors for resolving UV spectral signatures. Sci Adv. 2023 Nov 3;9(44):eadk3860. doi: 10.1126/sciadv.adk3860. Epub 2023 Nov 3. PMID 37922355